CLINICAL TRIAL: NCT05760053
Title: Toripalimab Plus Etoposide and Platinum-based Chemotherapy in First-line Treatment of Locally Advanced or Metastatic Genitourinary Small Cell Carcinoma：A Multicenter, Prospective, Open Label, Single-arm, Phase II Study
Brief Title: Toripalimab Plus Etoposide and Platinum-based Chemotherapy for Genitourinary Small Cell Carcinoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Shi Yanxia, Principal Investigator, Professor, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: B2023-013-01
Record Dates: First submitted 2023-02-18; First posted 2023-03-08 (Actual); Last update posted 2023-03-08 (Actual); Status verified 2023-03

CONDITIONS: Toripalimab; First-line Treatment
Keywords: Genitourinary small cell carcinoma; Carboplatin; Etoposide; Cisplatin
MeSH Terms: interventions — Etoposide; Cisplatin; Carboplatin

STUDY DESIGN:
Intervention Model Description: A multicenter, prospective, open label, single-arm, phase II study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- EP/EC+PD-1 (Experimental): Toripalimab 240mg D1 of each 21-day cycle IV drip; Etoposide 100mg/m2 D1-3 of each 21-day cycle IV drip; Cisplatin 25mg/m2 D1-3 of each 21-day cycle IV drip; Carboplatin AUC 5 D1 of each 21-day cycle IV drip;
  Interventions: Drug: EP/EC+PD-1

INTERVENTIONS:
Drug: EP/EC+PD-1 — Toripalimab 240 mg, administered on the first day of each cycle, and a cycle of administration every 3 weeks. Etoposide 100mg/m2, d1-3, cisplatin 25mg/m2, d1-3 or carboplatin AUC=5 d1, administered on the first day of each cycle, a cycle of administration every 3 weeks. Toripalimab combined with etoposide and cisplatin/carboplatin was used for 4 to 6 courses of treatment.
  Other Names: Etoposide, Cisplatin or Carboplatin, plus Toripalimab

SUMMARY:
This study is a prospective, multicenter, open-label, single-arm phase II clinical trial. A single-arm experimental group of toripalimab, etoposide, and cisplatin/carboplatin was designed to evaluate its efficacy and safety in small cell carcinoma of the urinary system.

DETAILED DESCRIPTION:
This study focuses on patients with locally advanced/metastatic genitourinary small cell carcinoma (small cell carcinoma originating in the kidney, ureter, bladder, urethra, and prostate), and it aims to explore the efficacy and safety of toripalimab combined with EP or EC.

After meeting the enrollment conditions, they received combination therapy: toripalimab 240 mg, administered on the first day of each cycle, and a cycle of administration every 3 weeks. Etoposide 100mg/m2, d1-3, cisplatin 25mg/m2, d1-3 or carboplatin AUC=5 d1, administered on the first day of each cycle, a cycle of administration every 3 weeks. Toripalimab combined with etoposide and cisplatin/carboplatin was used for 4 to 6 courses of treatment. Evaluate the curative effect with imaging every 2 courses. If there is an opportunity for local treatment after chemotherapy, participate in multidisciplinary discussions to decide the next step of treatment. For patients who can be treated with local treatment (surgery, radiotherapy) after treatment, the investigator will receive maintenance treatment with toripalimab 240 mg/time, every 21 days, until the disease progresses or unacceptable toxicity occurs. If the curative effect evaluation of the patient is complete remission (CR), partial remission (PR) or stable disease (SD) after 4 to 6 courses of treatment, maintenance therapy with toripalimab 240mg/time, every 21 days, until the disease progression or intolerable toxicity. The maximum duration of maintenance treatment is 2 years. Subjects who finished treatment entered the follow-up period and received safety follow-up and survival follow-up.

ELIGIBILITY:
Inclusion Criteria:

1. Participate voluntarily and sign the informed consent;
2. Age ≥ 18 years old;
3. Life expectancy ≥ 3 months;
4. Physical condition score ECOG 0-2;
5. Pathologically diagnosed as genitourinary small cell carcinoma (recommended central consultation for difficult pathology), including small cell carcinoma primary in the kidney, ureter, bladder, urethra, and prostate. The stage is locally advanced or advanced (stage IIIA or above, that is, cT3 or above N0 M0, or cT1-4a N1-3 M0, or cT4b any N M0, or any T any N M1), or the investigator judges that local treatment is not suitable for the time being (surgery, radiotherapy) patients.
6. Patients whose pathology is mixed small cell carcinoma can be included, and the small cell carcinoma component is ≥50%.
7. Have not received systemic treatment before, or the time interval from the last adjuvant treatment is more than 6 months;
8. There are measurable or/and evaluable lesions (non-radiotherapy target areas) (lesion evaluation according to Recist1.1 standard);
9. No serious organ (main organs: heart, lung, liver, kidney) dysfunction (refer to the respective standards);
10. Blood routine indicators: white blood cell (WBC) ≥ 3 × 109/L; absolute neutrophil count (ANC) ≥ 1.5 × 109/L; platelet (PLT) ≥ 100 × 109/L; hemoglobin (Hgb) ≥ 8g /dL;
11. Blood biochemical indicators: AST (SGOT), ALT (SGPT) ≤ 2.5 × upper limit of normal value (ULN) (in the case of no liver invasion) or ≤ 5 × upper limit of normal value (ULN) (in the case of liver invasion ); total bilirubin (TBIL) ≤ ULN; serum creatinine clearance calculated according to the CG formula > 30 mL/min
12. Coagulation function: prothrombin time (PT), international normalized ratio (INR) ≤ 1.5 × ULN (unless warfarin is being used for anticoagulation);
13. Able to comply with the research visit plan and other program requirements;
14. All patients of childbearing age must agree to take effective contraceptive measures during the study period and within 6 months of stopping treatment, and the urine pregnancy test of female patients of childbearing age must be negative before treatment.

Exclusion Criteria:

1. Received treatment for small cell carcinoma of the urinary system within 2 weeks before enrollment.
2. Once diagnosed with prostate adenocarcinoma, received endocrine therapy (such as enzalutamide, apalutamide, abiraterone, etc.) and chemotherapy (docetaxel) for prostate adenocarcinoma, and is currently considering neuroendocrine differentiation of prostate cancer.
3. Mixed small cell carcinoma, in which the small cell carcinoma component is less than 50%.
4. Medical history and comorbidities:

(1) Anti-tumor vaccine or cellular immunotherapy has been used before the first dose of the study drug; (2) Previously received systemic therapy for metastatic lesions; (3) The patient is participating in other interventional clinical studies or less than 4 weeks before the end of the previous clinical study; (4) Those who have been less than 4 weeks away from the last anti-tumor treatment (radiotherapy, chemotherapy, targeted therapy, immunotherapy or local-regional treatment). The adverse reactions related to anti-tumor treatment (except hair loss) after the previous systemic anti-tumor treatment have not recovered to NCI-CTC AE≤level 1; (5) Live vaccines have been vaccinated within 4 weeks before administration of the study drug. Inactivated virus vaccines for seasonal influenza and injection are allowed, but attenuated live influenza vaccines for intranasal administration are not allowed; (6) The subject has any active, known or suspected autoimmune disease. Subjects who are in a stable state and do not require systemic immunosuppressant therapy are allowed to be enrolled; (7) Subjects who required systemic treatment with corticosteroids (>10 mg/day of prednisone or equivalent doses of other glucocorticoids) or other immunosuppressants within 14 days before the first dose of study drug. Steroid replacement with inhaled or topical steroids and curative doses of prednisone at doses > 10 mg/day is permitted in the absence of active autoimmune disease; (8) Patients with a known history of interstitial pneumonia or highly suspected interstitial pneumonia; or patients who may interfere with the detection or treatment of suspected drug-related pulmonary toxicity; (9) Other active malignant tumors that require simultaneous treatment; (10) Has a history of malignant tumors. Patients with basal cell carcinoma of the skin, superficial bladder cancer, squamous cell carcinoma of the skin, or cervical carcinoma in situ who underwent potentially curative therapy and had no disease recurrence within 5 years from the end of treatment were excluded; (11) Known history of organ transplantation and allogeneic hematopoietic stem cell transplantation;(12) Subjects who have undergone major surgery or severe trauma have less than 14 days before enrollment; (13) Patients with active pulmonary tuberculosis should be excluded. Patients suspected of having active pulmonary tuberculosis should be checked for chest X-ray, sputum, and ruled out by clinical symptoms and signs. Patients with a history of active tuberculosis infection within the previous 1 year, even if treated, should be excluded; patients with a history of active tuberculosis infection more than 1 year ago should also be excluded. Unless it is proven that the duration and type of antituberculosis treatment previously used was appropriate; (14) Severe acute or chronic infection requiring systemic therapy； (15) Heart failure (New York Heart Association Class III or IV) despite appropriate medical therapy. Patients with poorly controlled coronary artery disease or poorly controlled arrhythmia, or a history of myocardial infarction within 6 months prior to screening.

5. Neutrophil count <1.0×109/L, or hemoglobin <80g/L, or platelet count <90×109/L. Hepatic insufficiency not related to tumor (transaminase more than 3 times the upper limit of normal value and/or blood bilirubin greater than 2.0mg/dl). Renal insufficiency not related to tumor (serum creatinine clearance <30 mL/min calculated according to the CG formula).

6. Known history of positive human immunodeficiency virus (HIV) or known acquired immunodeficiency syndrome (AIDS).

7. Untreated active hepatitis (hepatitis B: HBsAg positive and HBV DNA ≥ 500IU/mL; hepatitis C: HCV RNA positive and abnormal liver function); co-infected with hepatitis B and C.

8. Allergy to any study drug. 9. Pregnant and breastfeeding women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Estimated)
Dates: Start 2023-02-18 (Actual); Primary Completion 2025-02-18 (Estimated); Study Completion 2026-02-18 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) | Within approximately 36 months
  Progression-free survival (PFS) is defined as the time from the date of the first dose to the earlier of the dates of the first objective documentation of radiographic progressive disease (PD) or death due to any cause.

SECONDARY OUTCOMES:
Complete Response Rate (CRR) | Within approximately 36 months
  Percentage of participants with response reported as complete response
Duration of Response (DOR) | Within approximately 36 months
  Duration of response was defined as the time interval between the date of first documentation of objective response (CR or PR) and the date of the first objective documentation of disease progression or death due to any cause.
Objective Response Rate (ORR) | Within approximately 36 months
  The number of participants with objective response is assessed every six weeks from Cycle 1 Day 1 through discontinuation of treatment. Objective response rate (ORR) was defined as the proportion of participants who achieved a best overall response of complete response or partial response based on local radiologists/investigators' tumor assessments.
Overall Survival (OS) | Within approximately 36 months
  Overall survival (OS) is defined as the time from the date of first dose to the date of death from any cause.
Incidence of Treatment-related Adverse Events | Within approximately 36 months
  Incidence of Treatment-related Adverse Events as assessed by the National Cancer Institute's Common Terminology Criteria for Adverse Events (CTCAE, Version 5.0).

CONTACTS AND LOCATIONS:
Overall Officials: Yanxia Shi, Principal Investigator — Sun Yat-sen University
Locations (1):
- Sun Yat-sen University cancer center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-10-15): https://cdn.clinicaltrials.gov/large-docs/53/NCT05760053/Prot_SAP_000.pdf
  • Informed Consent Form (2022-10-15): https://cdn.clinicaltrials.gov/large-docs/53/NCT05760053/ICF_001.pdf